CLINICAL TRIAL: NCT05892315
Title: Timing of Re-evaluation After Steps I-II of Periodontal Therapy: a Randomized Clinical Trial
Brief Title: Timing of Re-evaluation After Steps I-II of Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTurin3
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Dental Scaling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated subgingival instrumentation (Experimental): Conventional staged debridement (CSD) according to the severity of periodontitis in 2 to 4 appointments at day 0, 7, 14 and 21. Re-instrumentation at 6 weeks and 3 months after completion of step I-II.
  Interventions: Procedure: Repeated subgingival instrumentation
- Supragingival instrumentation (Active Comparator): Conventional staged debridement (CSD) according to the severity of periodontitis in 2 to 4 appointments at day 0, 7, 14 and 21. Only supragingival instrumentation at 6 weeks and 3 months after completion of step I-II.
  Interventions: Procedure: Supragingival scaling

INTERVENTIONS:
Procedure: Repeated subgingival instrumentation — Supragingival scaling will be performed at sites with plaque and subgingival scaling will be performed by the use of manual and ultrasonic instruments at pockets ≥ 4 mm with bleeding. Oral hygiene instructions will be reinforced. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.
  Arms: Repeated subgingival instrumentation
Procedure: Supragingival scaling — Supragingival scaling will be performed at sites with plaque. Oral hygiene instructions will be reinforced. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.
  Arms: Supragingival instrumentation

SUMMARY:
Literature on non surgical periodontal therapy (NSPT) shows lack of clarity in reporting information on re-evaluation timing and clinical response. If the re-evaluation was done shortly after NSPT, this is also likely to have an influence on the surgical treatment plan. The aim of this randomized clinical trial is to investigate the effect of re-evaluation timing at 1-3-6 months after NSPT in terms of pocket closure, probing pocket depth reduction, comprehensive treatment plan, and costs for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage III-IV
* Full-mouth plaque score (FMPS) < 25% at the 1-month re-evaluation
* Full-mouth bleeding score (FMBS) < 25% at the 1-month re-evaluation
* Signed informed consent

Exclusion criteria:

* Age < 18 yo
* Pregnancy or lactation
* Heavy smokers (>10 die)
* Conditions or diseases influencing periodontal healing
* Patients that cannot complete the 6 months follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-06-11 (Estimated); Study Completion 2024-12-11 (Estimated)

PRIMARY OUTCOMES:
Change in treatment success % (0 - 100 % with higher percentage indicating better status) | Baseline, 1 month, 3 months and 6 months after the completion of the therapy.
  Percentage of pockets ≥ 4 mm with bleeding that converted to ≤ 3 mm or ≤4 mm without bleeding at the completion of non-surgical periodontal therapy

SECONDARY OUTCOMES:
Change in Full Mouth Plaque Score (FMPS%) (0 - 100 % with higher percentage indicating worse status) | Baseline, 1 month, 3 months and 6 months after the completion of the therapy.
  Percentage of full mouth plaque score considering 6 sited for each tooth.
Change in Probing Pocket Depth (PD) (0 - 15 mm with higher values indicating worse outcomes). | Baseline, 1 month, 3 months and 6 months after the completion of the therapy.
  The distance between the cementoenamel junction (CEJ) and the base of the pocket.
Change in Clinical Attachment Level (CAL) (0 - 15 mm with higher values indicating worse outcomes). | Baseline, 1 month, 3 months and 6 months after the completion of the therapy.
  The sum of Probing pocket depth (PD, mm) and Recession (Rec, mm).

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy